CLINICAL TRIAL: NCT02712515
Title: The Motor Network in Essential Tremor: Mechanisms of Therapy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201600172-N; 03UH3NS095553 (Other Grant/Funding Number: National Institute of Neurological Disorders and Stroke)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2025-08

CONDITIONS: Essential Tremor; Parkinson's Disease
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Essential tremor: Participants in this group will be undergoing deep brain stimulation implantation surgery as part of the standard of care. In addition, the Ad-Tech Medical Instrumentation Corp. device will be used to test responses with wireless sensors placed on the participant's arms, which can record EMG activity. Brain signals will be recorded using the clinical FHC Guideline 4000+ system and/or Medtronic RC+S devices, which are capable of recording during stimulation.
  Interventions: Procedure: Deep brain stimulation implantation surgery; Device: Ad-Tech Medical Instrumentation Corp. electrodes/subdural strips; Device: FHC Guideline 4000+ system and/or Medtronic RC+S
- Parkinson's disease and dystonia: Participants in this group with Parkinson's disease and/or dystonia will be undergoing deep brain stimulation implantation surgery as part of the standard of care. In addition, the Ad-Tech Medical Instrumentation Corp. device will be used to test responses with wireless sensors placed on the participant's arms, which can record EMG activity. Brain signals will be recorded using the clinical FHC Guideline 4000+ system and/or Medtronic RC+S devices, which are capable of recording during stimulation.
  Interventions: Procedure: Deep brain stimulation implantation surgery; Device: Ad-Tech Medical Instrumentation Corp. electrodes/subdural strips; Device: FHC Guideline 4000+ system and/or Medtronic RC+S

INTERVENTIONS:
Procedure: Deep brain stimulation implantation surgery — Deep brain stimulation is a neuromodulatory therapy in which electrodes are implanted in deep brain structures. Electrical pulses are delivered through these electrodes to suppress pathological activity that are causing the symptoms of essential tremor or Parkinson's disease.
Device: Ad-Tech Medical Instrumentation Corp. electrodes/subdural strips — Ad-Tech Medical Instrumentation Corp. electrodes are intraoperative monitoring subdural strips will be placed on the surface of the cortex (non-penetrating).
  Other Names: Ad-tech intraoperative monitoring subdural strips
Device: FHC Guideline 4000+ system and/or Medtronic RC+S — Brain signals will be recorded using the clinical Participants in this group with Parkinson's disease will be undergoing deep brain stimulation implantation surgery as part of the standard of care. In addition, the Ad-Tech Medical Instrumentation Corp. device will be used to test responses with wireless sensors placed on the participant's arms, which can record EMG activity. Brain signals will be recorded using the clinical FHC Guideline 4000+ system and/or Medtronic RC+S devices, which are capable of recording during stimulation.

SUMMARY:
Essential tremor (ET) is among the most common movement disorders, and is the most prevalent tremor disorder. It is a progressive, degenerative brain disorder that results in increasingly debilitating tremor, and afflicts an estimated 7 million people in the US (2.2% of the population) and estimates from population studies worldwide range from 0.4% to 6.3%. ET is directly linked to progressive functional impairment, social embarrassment, and even depression. Intention (kinetic) tremor of the arms occurs in approximately half of ET patients, and is typically a slow tremor (~5-10Hz) that occurs at the end of a purposeful movement, and is insidiously progressive over many years. Based on direct and indirect neurophysiological studies, it has been suggested that a pathological synchronous oscillation in a neuronal network involving the ventral intermediate nucleus (Vim) of the thalamus, the premotor (PM), primary motor (M1) cortices, and the cerebellum, may result in the production of ET. In spite of the numerous therapeutic modalities available, 65% of those suffering from upper limb tremor report serious difficulties during their daily lives. Deep brain stimulation (DBS) has emerged as an effective treatment option for those suffering from medically refractory ET. The accepted target for ET DBS therapy is the Vim thalamus. Vim projects to PM, M1, and supplementary motor areas (SMA) and receives afferents from the ipsilateral cerebellum. Moreover, electrophysiological recordings from Vim during stereotactic surgery have identified "tremor cells" that synchronously discharge with oscillatory muscle activity during tremor. Clinical and computational findings indicate that DBS suppresses tremor by masking these "burst driver" inputs to the thalamus. The overall goal is to investigate the neural signatures of tremor generation in the thalamocortical network by recording data during DBS implantation surgery. Investigators will record data from the macroelectrode implanted in the Vim for DBS therapy, and through an additional 6-contact subdural cortical strip that will be placed on the hand motor cortical area temporarily through the same burr hole opened for the implantation of the DBS electrode.

DETAILED DESCRIPTION:
The research study goal is to advance the understanding of the mechanisms for essential tremor through brain recordings. The investigators will collect brain signals in persons with essential tremor undergoing neurosurgical treatment (deep brain stimulation implantation). By recording from the implanted electrodes for deep brain stimulation along with two other non-invasive intraoperative monitoring electrodes, the origins of tremor will be studied in the human motor network. Moreover, by performing recordings during deep brain stimulation delivery, the mechanisms in which deep brain stimulation modulates this network to suppress tremor will be investigated.

During the standard of care DBS procedure neural recordings are performed as the participant is in a reclined position on the operating table. In addition to neural recordings it is standard to ask the patient to move their arms and legs during the procedure. An additional intraoperative monitoring subdural electrode strip, used in epilepsy and tumor surgeries to perform functional mapping, will be placed by the neurosurgeon after the DBS electrode is placed per the clinical need of the patient. In addition, the Ad-Tech Medical Instrumentation Corp. device will be used to test responses with wireless sensors placed on the participant's arms, which can record electromyogram (EMG) activity. Brain signals will be recorded using the clinical NeuroOmega system Medtronic RC+S, which are devices capable of recording during stimulation. This additional testing will add approximately 30-45 minutes to the surgical time. The Medtronic RC+S stimulator will not be implanted in these subjects, and will not used as a therapy. No interventions are compared against any controls for this study.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical patient populations with essential tremor (main cohort) and Parkinson's disease (control cohort)

Exclusion Criteria:

* Non surgical candidates

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgical patient populations with essential tremor (main cohort) and Parkinson's disease (control cohort)
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Brain signals between the groups | intraoperative
  FHC Guideline 4000+ system or Medtronic devices will be connected to Ad-Tech Medical Instrumentation Corp. electrodes and deep brain electrodes to measure brain signals between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gunduz, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided